CLINICAL TRIAL: NCT04992169
Title: Clinicianless Training in Autism Treatment: An Adaptive Online Parent Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Santa Barbara (Other)
Responsible Party: Principal Investigator, Ty Vernon, Associate Professor, University of California, Santa Barbara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-21-0034
Record Dates: First submitted 2021-06-18; First posted 2021-08-05 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder; Parents
Keywords: Autism; Treatment; Intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial with two arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant families will be randomly assigned by the smartphone app to one arm or the other. While caregivers are not directly notified of their group/arm assignment, their participation in arm-specific app-tasks may help them determine which arm they are assigned to. Investigators and outcomes assessors remain masked to condition until data collection and analysis is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smartphone App with Video Self-Scoring Functionality (Experimental): In this condition, after parents video-record their delivery of the intervention, they watch their video and are taught to score their own performance/fidelity through question prompts built into the app. When they are finished, the app will offer feedback and follow-up lessons based on the PRT strategies they have not demonstrated consistently.
  Interventions: Behavioral: Smartphone-App Parent Training in Pivotal Response Treatment
- Smartphone App without Video Self-Scoring Functionality (Experimental): In this condition, after parents video-record their delivery of the intervention, they watch their own video but do not score their performance.
  Interventions: Behavioral: Smartphone-App Parent Training in Pivotal Response Treatment

INTERVENTIONS:
Behavioral: Smartphone-App Parent Training in Pivotal Response Treatment — Parents are trained in Pivotal Response Treatment, Pivotal Response Treatment is a well-known, scientifically supported treatment that focuses on using child motivation, play-based lessons, and parent involvement to target the language skills and social engagement of children with autism. The core smartphone app will offer eight interactive lessons in PRT, consisting of video examples, slides, and brief quizzes.

SUMMARY:
This project will examine the feasibility, acceptability, and preliminary efficacy of using a smartphone app-based parent training program focused on early autism intervention strategies.

DETAILED DESCRIPTION:
Despite scientific advances in treatment for autism spectrum disorder (ASD), most families across the United States do not have access to high quality autism services, let alone the best autism treatment models available. There are a number of reasons for this concerning reality, including the limited number of trained autism clinicians around the country, the rising cost of services, geographic distance from autism service providers, and difficulties in being able to effectively and efficiently train a large number of people in the latest treatment models.

This proposed project focuses on the Department of Defense Autism Research Program - Clinical Translational Research Award Area of Interests focused on Dissemination/Implementation of Clinically Validated Interventions and Behavioral Therapies for ASD Core Symptoms. These areas focus on effective strategies for taking what works (in this case, highly effective autism treatments shown to improve social communication and motivation in children with autism) and spreading or distributing these treatments so that they can benefit a much larger portion of the population. This is important, because a highly effective treatment is of little use if only people in a few areas can benefit from its effect, while the rest of the nation continues to use outdated, less effective strategies.

To accomplish the goal of distributing a highly effective intervention to the general public, this proposed study will take advantage of the wide-spread use of smartphones nationwide. This study proposes to develop and evaluate smartphone apps as a way to train parents of young children with ASD in an autism treatment model known as Pivotal Response Treatment (PRT). Families will be recruited nationwide to participate in this trial.

Pivotal Response Treatment is a well-known, scientifically supported treatment that focuses on using child motivation, play-based lessons, and parent involvement to target the language skills and social engagement of children with ASD. The core smartphone app will offer eight interactive lessons in PRT, consisting of video examples, slides, and brief quizzes. After each lesson, parents will be asked to record a brief video of themselves using PRT with their child, which is submitted within the app to the research team so that they can monitor their mastery of the strategies over time. The investigators will also ask parents to complete autism-related and developmental surveys before and after participation so that the research team can monitor how their child is improving.

Ultimately, the objective of this trial is to develop and test smartphone apps to deliver a highly effective autism intervention to families nationwide. The use of this technology will ensure that families can access gold standard autism treatment regardless of their geographic location, work schedules, or financial background. If successful, the investigators plan to conduct an even larger nationwide study and ultimately make the app available in smartphone app stores so that families everywhere can train themselves in this treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autism spectrum disorder
* Parent endorsements of significant language delay
* Between the ages of 1.0 and 4.5 years (12 and 54 months)
* Parents willing to complete intake and follow-up assessments, complete the eight weekly PRT lessons, record and submit parent-child PRT videos, and review these videos on a weekly basis.
* Access to an internet connection and an iOS smartphone or tablet that can supports the app and records video.

Exclusion Criteria:

* Significant medical conditions, seizures, and mental health concerns
* Non-English speaking
* Prior parent training in PRT or similar Naturalistic Developmental Behavioral Intervention

Ages: 12 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Parent Fidelity of Implementation of Pivotal Response Treatment (PRT) during Behaviorally Coded Parent-Child Intervention Videos at 8 weeks, 16 weeks | Baseline, 8 weeks (intervention completion), 16 weeks (follow-up)
  Parent participants will record and submit a five-minute video of themselves using the PRT intervention strategies with their child using the clinical trial's smartphone app. Trained research assistants will behaviorally score each video using computer-based behavioral coding software (Noldus Observer XT) on a trial-by-trial basis for the presence or absence of each PRT intervention component, which include the use of: child choice, child attention, clear opportunities, contingent reinforcement, reinforcement of child response attempts, a balance of maintenance and acquisition tasks, and task variation. Total uses of these components will be divided by total uses + absences of these components to yield a percentage. The mean percentage of all components will be used as the primary outcome, with a range of 0% to 100% use of the PRT components.

SECONDARY OUTCOMES:
Change from Baseline in Frequency of Child Vocalizations/Word Use during Behaviorally Coded Parent-Child Intervention Videos at 8 weeks, 16 weeks. | Baseline, 8 weeks (intervention completion), 16 weeks (follow-up)
  Parent participants will record and submit a five-minute video of themselves using the PRT intervention strategies with their child using the clinical trial's smartphone app. Trained research assistants will behaviorally score each video using computer-based behavioral coding software (Noldus Observer XT) on a continuous basis for the total frequency of child vocalizations and word use (both prompted and unprompted/spontaneous). The minimum number of vocalizations/words is 0 (no vocalizations or spoken words) and there is technically no maximum (although this is limited by the 5-minute duration of the video probe).
Change from Baseline in Percentage of Child Positive Affect during Behaviorally Coded Parent-Child Intervention Videos at 8 weeks, 16 weeks. | Baseline, 8 weeks (intervention completion), 16 weeks (follow-up)
  Parent participants will record and submit a five-minute video of themselves using the PRT intervention strategies with their child using the clinical trial's smartphone app. Trained research assistants will behaviorally score each video using computer-based behavioral coding software (Noldus Observer XT) on a continuous basis for the total duration of child positive affect (i.e. directed positive facial expressions - observable smiling and laughter). The minimum percentage is 0% (no positive affect) and the maximum is 100% (constant presence of positive affect).
Change from Baseline in MacArthur-Bates Communicative Development Inventory (CDI), Level I Short Form (Total Score) at 16 weeks | Baseline, 16 weeks (follow-up)
  The MacArthur-Bates CDI (Fenson et al., 2000) is a caregiver-reported measure of child expressive vocabulary use. Parents will complete a digital version of the CDI to obtain information on reported word usage and understanding.
Change from Baseline in Vineland Adaptive Behavior Scales, Third Edition (Standard Score on Communication Domain) at 16 weeks | Baseline, 16 weeks (follow-up)
  The Vineland-III (Sparrow et al., 2016) is a caregiver-completed measure of adaptive functioning in children. Parents will complete a digital version of the Communication Domain of the Vineland-III Parent/Caregiver Rating Form. Item responses are converted to Standard Scores with a mean of 100 and a Standard Deviation of 15.
Change from Baseline in Vineland Adaptive Behavior Scales, Third Edition (Standard Score on Socialization Domain) at 16 weeks | Baseline, 16 weeks (follow-up)
  The Vineland-III (Sparrow et al., 2016) is a caregiver-completed measure of adaptive functioning in children. Parents will complete a digital version of the Socialization Domain of the Vineland-III Parent/Caregiver Rating Form. Item responses are converted to Standard Scores with a mean of 100 and a Standard Deviation of 15.
Change from Baseline in Social Responsiveness Scale, Second Edition (SRS-2; Total T-Score) at 16 weeks | Baseline, 16 weeks (follow-up)
  The SRS-2 (Constantino & Gruber, 2007) is a caregiver-completed measure of a child's autism symptom severity. Parents will complete a digital version of the Toddler SRS-2. Item responses are converted to a SRS-2 T-score with a mean of 50 and a Standard Deviation of 10.

OTHER OUTCOMES:
Change from Baseline in Percentage of Child Eye Contact during Behaviorally Coded Parent-Child Intervention Videos at 8 weeks, 16 weeks. | Baseline, 8 weeks (intervention completion), 16 weeks (follow-up)
  Parent participants will record and submit a five-minute video of themselves using the PRT intervention strategies with their child using the clinical trial's smartphone app. Trained research assistants will behaviorally score each video using computer-based behavioral coding software (Noldus Observer XT) on a continuous basis for the total frequency and duration of child eye contact (i.e. child gazing in the direction of the caregiver's head). The minimum percentage is 0% (no eye contact) and the maximum is 100% (constant eye contact).
Scale of Treatment Perceptions (Total Score) | 8 weeks
  The Scale of Treatment Perceptions (STP; Berger, et al., 2016) assesses parents' satisfaction with intervention using the mean of survey items with 1-7 Likert rating scale, with higher scores indicating higher levels of satisfaction (better outcome).
Parent Adherence to Treatment and Competence Measure | 8 weeks
  The PATC is a six-item self-report adherence-to-treatment and competence measure (PATC; Kasari et al., 2010) will be administered to parents once they complete the app program. The measure consists of four items concerning adherence to treatment protocol: (1) made time to carry out the learned strategies, (2) found it complex to carry out the learned strategies, (3) thought it natural to carry out the learned strategies, and (4) made an effort to carry out the learned strategies. The PATC also includes two items concerning parental competence: (1) was confident carrying out the learned strategies, and (2) was comfortable carrying out the learned strategies. All items consist of a series of ratings on a 1-5 Likert rating scale, with higher scores indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ty Vernon, Principal Investigator — University of California, Santa Barbara
Locations (1):
- University of California, Santa Barbara, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: Yes
As part of the informed consent process, participants will consent to allow their deidentified data to be shared with National Database for Autism Research (NDAR).
Supporting Information: Study Protocol, SAP
Time Frame: Participant trial data will be submitted in months 23-24 of the trial.

DOCUMENTS (3):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04992169/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04992169/SAP_001.pdf
  • Informed Consent Form (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04992169/ICF_002.pdf